CLINICAL TRIAL: NCT01204125
Title: Randomized, Open-label, Phase 2 Study of the Efficacy and Safety of Weekly Paclitaxel Single-agent and Two Different Regimens of the PARP-1 Inhibitor SAR240550 (BSI-201) in Combination With Weekly Paclitaxel, as Neoadjuvant Therapy in Patients With Stage II-IIIA Triple Negative Breast Cancer (TNBC)
Brief Title: Two Regimens of SAR240550/Weekly Paclitaxel and Paclitaxel Alone as Neoadjuvant Therapy in Triple Negative Breast Cancer Patients
Acronym: SOLTI NEOPARP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD11419; 2010-018960-17 (EudraCT Number)
Record Dates: First submitted 2010-09-13; First posted 2010-09-17 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Paclitaxel; iniparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SAR240550 twice weekly/ paclitaxel weekly (Experimental): SAR240550 will be administered at the dose of 5.6mg/kg as a 60-min intravenous (IV) infusion. Patients will receive SAR240550 infusions twice weekly (day 1 and day 4; total dose of 11.2mg/kg per week) and paclitaxel weekly as a 60-min IV infusion (day 1; dose of 80mg/m2).
  Interventions: Drug: Iniparib (SAR2405550 -BSI-201)
- SAR240550 weekly/ paclitaxel weekly (Experimental): SAR240550 will be administered at the dose of 11.2 mg/kg as a 60-min intravenous (IV) infusion. Patients will receive SAR240550 infusions once weekly (day 1; total dose of 11.2mg/kg per week) and paclitaxel weekly as a 60-min IV infusion (day 1; dose of 80mg/m2).
  Interventions: Drug: Iniparib (SAR2405550 -BSI-201)
- Paclitaxel alone (Active Comparator): Paclitaxel will be administered at the dose of 80mg/m2 as a 60-min IV infusion. Patients will receive weekly (day 1) paclitaxel infusions.
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: paclitaxel — Pharmaceutical form:solution for infusion
  Route of administration: intravenous
  Arms: Paclitaxel alone
Drug: Iniparib (SAR2405550 -BSI-201) — Pharmaceutical form : solution for infusion
  Route of administration :Intravenous
  Arms: SAR240550 twice weekly/ paclitaxel weekly; SAR240550 weekly/ paclitaxel weekly

SUMMARY:
Primary Objective:

- to assess the pathological Complete Response (pCR) rate in the breast of patients treated in following combinations: SAR240550 twice-weekly + weekly paclitaxel, SAR240550 weekly+ weekly paclitaxel, and weekly paclitaxel single agent as calibrator.

Secondary objectives are:

* pCR rate in the breast and axilla,
* Radiological/clinical objective response rate (ORR), breast conservation rate, disease free survival (DFS), and overall survival (OS), in each treatment arm,
* Safety profiles of study combinations and of the single agent reference treatment,
* Molecular characteristics of the tumor tissue and peripheral blood mononuclear cells (PBMC) and any correlation between the biological activity of the study treatment and the disease outcome.

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

DETAILED DESCRIPTION:
Active study treatment will be given either as twice weekly administration (Day 1 and Day 4) or as weekly administration (Day 1) for a maximum of 24 infusions for Arm A and for a maximum of 12 infusions for Arm B. In all study arms, treatment will be given until definitive surgery, the first sign of disease progression, unacceptable toxicity or withdrawal of patient consent.

Definitive surgery will be performed within 2 to 4 weeks after the last dose of study treatment.

Patients who complete all the study treatment or who withdraw consent or experience intolerable toxicity will undergo surgery according to local practices.

The cut-off date for the primary analyses will be 30 days after the last study treatment administration or the date of the definitive surgery, whichever comes last.

The maximum follow up for each individual patient will be until death or 5 years after the definitive surgery date whatever happens first.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed Stage II-IIIA invasive breast cancer eligible for definitive surgery and Estrogen Receptor (ER)-negative, Progesterone receptor (PgR)-negative and Human epidermal growth factor receptor 2 (HER2) non-overexpressing by Immunohistochemistry (IHC) (0+, 1+) or fluorescence in situ hybridization (FISH negative, ratio <1.8) or IHC (2+, 3+) /FISH-negative.
* The primary tumor must be > 2cm in diameter measured by physical examination and mammography (mandatory) plus either echography or Magnetic Resonance Imaging (MRI)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate bone marrow reserve
* Adequate liver and renal function.
* Age > or = 18 years

Exclusion criteria:

* Any prior treatment for primary breast cancer.
* Bilateral or multicentric breast cancer.
* Other primary tumors within the previous 5 years, except for adequately controlled limited basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Pre-existing peripheral neuropathy grade > or = 2 as per National Cancer Institute Common Toxicity Criteria for Adverse Event (NCI CTCAE) at randomization.
* Any history of medical (e.g., cardiovascular, uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled infection) or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, may increase the risks associated with the study participation or administration of the investigational products, or that may interfere with the interpretation of the results
* Pregnancy or breastfeeding women.
* Women of childbearing potential (<2 years after the last menstruation) not using effective, non-hormonal means of contraception during the study and for a period of 6 months following the last administration of study drug.
* Requirement for radiation therapy concurrent with study anticancer treatment. Patients who require breast or chest wall radiation therapy after surgery are eligible.
* Known hypersensitivity to any of the study drugs or excipients

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate defined as the complete absence of invasive carcinoma on histological examination of the breast at the time of definitive surgery and confirmed by blinded centralized review | at the time of definitive surgery

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) rate in the breast and axilla | at the time of definitive surgery
Objective Response Rate(ORR) defined in the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) as complete response rate + partial response rate | at the time of definitive surgery
Breast conservation rate | at the time of definitive surgery
Disease Free Survival rate (DFS) | up to a maximum of 5 years after definitive surgery
Overall Survival (OS) | up to a maximum of 5 years after definitive surgery
Safety parameters (number of patients AE, SAE or AEPM) | up to a maximum of 5 years after definitive surgery
Molecular-biological testing | 2 or 3 timepoints during treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (25):
- France (6):
  - Investigational Site Number 250001, Besançon
  - Investigational Site Number 250004, Bordeaux
  - Investigational Site Number 250006, Bron
  - Investigational Site Number 250003, Paris
  - Investigational Site Number 250002, Toulouse
  - Investigational Site Number 250005, Villejuif
- Germany (4):
  - Investigational Site Number 276002, Cologne
  - Investigational Site Number 276003, Erlangen
  - Investigational Site Number 276004, Hamburg
  - Investigational Site Number 276001, Mönchengladbach
- Spain (15):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724009, Cáceres
  - Investigational Site Number 724013, Córdoba
  - Investigational Site Number 724006, Islas Baleares
  - Investigational Site Number 724012, Jaén
  - Investigational Site Number 724002, Lleida
  - Investigational Site Number 724005, Madrid
  - Investigational Site Number 724016, Madrid
  - Investigational Site Number 724007, Reus
  - Investigational Site Number 724018, Santiago de Compostela
  - Investigational Site Number 724017, Seville
  - Investigational Site Number 724010, Seville
  - Investigational Site Number 724003, Torrevieja
  - Investigational Site Number 724011, Valencia
  - Investigational Site Number 724015, Valencia

REFERENCES:
- [Derived] Llombart-Cussac A, Bermejo B, Villanueva C, Delaloge S, Morales S, Balmana J, Amillano K, Bonnefoi H, Casas A, Manso L, Roche H, Gonzalez-Santiago S, Gavila J, Sanchez-Rovira P, Di Cosimo S, Harbeck N, Charpentier E, Garcia-Ribas I, Radosevic-Robin N, Aura C, Baselga J. SOLTI NeoPARP: a phase II randomized study of two schedules of iniparib plus paclitaxel versus paclitaxel alone as neoadjuvant therapy in patients with triple-negative breast cancer. Breast Cancer Res Treat. 2015 Nov;154(2):351-7. doi: 10.1007/s10549-015-3616-8. Epub 2015 Nov 4. PMID 26536871